CLINICAL TRIAL: NCT02721303
Title: Appetite Regulation in Older-Aged Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1511
Record Dates: First submitted 2016-03-21; First posted 2016-03-29 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Obesity; Aging
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- obese older aged, aged 65-85, BMI 30-40 (Active Comparator): Older aged patients who are obese and between the ages of 65-85 with a BMI between 30-40.
  Interventions: Dietary Supplement: 3-day diet Run-in; Procedure: fMRI; Procedure: Intravenous catheter placed for blood draws
- normal weight older aged, aged 65-85, BMI 18-25 (Active Comparator): Older aged patients who are of normal weight and between the ages of 65-85 with a BMI between 18-25.
  Interventions: Dietary Supplement: 3-day diet Run-in; Procedure: fMRI; Procedure: Intravenous catheter placed for blood draws
- obese younger aged, aged 21-45, BMI 30-40 (Active Comparator): Younger aged patients who are obese and between the ages of 21-45 with a BMI between 30-40 .
  Interventions: Dietary Supplement: 3-day diet Run-in; Procedure: fMRI; Procedure: Intravenous catheter placed for blood draws

INTERVENTIONS:
Dietary Supplement: 3-day diet Run-in — Participants will be studied on one occasion after a 3-day diet run-in. This will be followed by a breakfast meal.
Procedure: fMRI — After a 3-day diet run-in, participants will undergo a functional magnetic resonance imaging procedure (fMRI). Repeat fMRI will be performed 30 minutes after the meal.
  Other Names: Functional Magnetic Resonance Imaging
Procedure: Intravenous catheter placed for blood draws — On the study day participants will present in the fasting state, have an intravenous catheter placed for blood draws and have baseline blood samples taken. Blood and appetite measures will be performed every half hour for 3 hours.
  Other Names: IV catheter

SUMMARY:
This study plans to learn more about how age and weight impact appetite and food intake. Specifically, this study is being done to see whether age and obesity impact appetite and the brain's response to food. In this study the investigators will be evaluating how participants brains respond to food images as well as your food-related behaviors and hormones. The investigators will be comparing older individuals aged 65 to 85 years who are normal weight compared to those who are obese. The Investigators will then compare older aged individuals to younger adults aged 21 to 45 years.

DETAILED DESCRIPTION:
In a cross sectional design participants will be studied on one occasion after a 3-day diet run-in. On the study day they will present in the fasting state, have an intravenous catheter placed for blood draws and have baseline blood samples taken and appetite measures performed. Participants will then undergo functional magnetic resonance imaging (fMRI). This will be followed by a breakfast meal. Blood and appetite measures will be performed every half hour for 3 hours. Repeat fMRI will be performed 30 minutes after the meal. After three hours participants will be offered a buffet style lunch and then will be done with the study visit.

ELIGIBILITY:
Inclusion Criteria:

* Older aged adults (O): 65-85
* Younger adults (Y): 21-45
* Obese (Ob): body mass index (BMI) 30-40
* Normal Weight (NW): BMI 18-25

Exclusion Criteria:

* Pregnancy;
* Advanced organ failure;
* Active cancer diagnosis;
* Uncontrolled hypertension or metabolic disorder;
* Cognitive impairment or psychiatric disease limiting ability to comply;
* Presently in an exercise or diet program;
* Recent weight loss of >5 lbs in past 6 mo.;
* Bariatric surgery;
* Use of any weight loss drugs;
* Use of any medication known to significantly affect appetite (anti-depressants are allowable);
* Present tobacco use;
* Use/abuse of substances of abuse including any marijuana use by history;
* Any contraindication to MRI;
* Claustrophobia;
* Body weight >300 lbs; and
* Inability to fit in MRI scanner.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
neuronal response to food images | 1 day
  fMRI of brain will be done in response to images of food

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Andre Cornier, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Univeristy of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No